CLINICAL TRIAL: NCT04019561
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Pharmacodynamic Effects of MEDI0382 in Obese Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)/ Non-Alcoholic Steatohepatitis (NASH)
Brief Title: A Study to Evaluate Safety and Pharmacodynamic Efficacy of 0382 in Obese Subjects With NAFLD/NASH.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5671C00002
Record Dates: First submitted 2019-06-24; First posted 2019-07-15 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-11

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Non-alcoholic Steatohepatitis (NASH)
Keywords: Non-alcoholic fatty liver disease; NAFLD; Non-alcoholic steatohepatitis; NASH; 0382
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MEDI0382 high dose (Experimental): MEDI0382 high dose administered subcutaneously
  Interventions: Drug: MEDI0382 high dose
- Placebo for MEDI0382 high dose (Placebo Comparator): Placebo for MEDI0382 high dose administered subcutaneously
  Interventions: Drug: Placebo for MEDI0382 high dose
- MEDI0382 low dose (Experimental): MEDI0382 low dose administered subcutaneoously
  Interventions: Drug: MEDI0382 low dose
- Placebo for MEDI0382 low dose (Placebo Comparator): Placebo for MEDI0382 low dose administered subcutaneously
  Interventions: Drug: Placebo for MEDI0382 low dose

INTERVENTIONS:
Drug: MEDI0382 high dose — MEDI0382 high dose administered subcutaneously
  Other Names: Cotadutide high dose
  Arms: MEDI0382 high dose
Drug: Placebo for MEDI0382 high dose — Placebo for MEDI0382 high dose administered subcutaneously
  Other Names: Placebo high dose
  Arms: Placebo for MEDI0382 high dose
Drug: MEDI0382 low dose — MEDI0382 low dose administered subcutaneously
  Other Names: Cotadutide low dose
  Arms: MEDI0382 low dose
Drug: Placebo for MEDI0382 low dose — Placebo for MEDI0382 low dose administered subcutaneously
  Other Names: Placebo low dose
  Arms: Placebo for MEDI0382 low dose

SUMMARY:
A Phase 2 study with 4 treatment groups of two differing doses and matched placebos designed to evaluate the safety (including hepatic safety), tolerability and pharmacodynamic effects of two dose levels of MEDI0382 in obese subjects with non-alcoholic fatty liver disease (NAFLD)/non-alcoholic steatohepatitis (NASH). The subjects will have biopsy-confirmed NAFLD/NASH with liver fibrosis stage F1, F2 or F3. Approximately 72 subjects will be randomized

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, study to evaluate the safety (including hepatic safety), tolerability and pharmacodynamic effects of two dose levels of MEDI0382 in obese subjects with non-alcoholic fatty liver disease (NAFLD)/non-alcoholic steatohepatitis (NASH). The subjects will have biopsy-confirmed NAFLD/NASH with liver fibrosis stage F1, F2 or F3. Approximately 72 subjects will be randomized across multiple study sites.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent (with the exception of consent for future genetic and non genetic research) prior to performing any study-specific procedures, including screening evaluations.
2. Subjects aged ≥ 18 years at the time of consent.
3. Body mass index ≥ 30 kg/m2 at screening.
4. HbA1c ≤ 9.5% (inclusive) at screening if T2DM present, managed by either diet and/or a stable dose of metformin, sodium-glucose co-transporter 2 (SGLT-2) inhibitors, sulphonylureas or acarbose (ie, no major dose adjustments in prior 3 months to screening).
5. Definitive NAFLD / NASH with NASH activity score (NAS) ≥ 4 with ≥ 1 in each component (i.e. steatosis, lobular inflammation and ballooning), as diagnosed by liver biopsy within 6 months of screening with liver fibrosis stage F1, F2 or F3. The number of subjects with F1 will be capped at 25% in the study.
6. Evidence of hepatic steatosis or liver fat (≥ 10%) by MRI.
7. Women of childbearing potential:

   1. Who are sexually active with a non-sterilized male partner must have used at least one highly effective method of contraception from screening, and must agree to continue using such precautions through to the end of the study. It is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.
   2. Must have a negative urine pregnancy test within 72 hours prior to the first dose of investigational product; and not be breastfeeding.

Exclusion Criteria:

1. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, put the subject at risk, influence the subject's ability to participate or affect the interpretation of the results of the study.
2. Liver disease of other etiologies (eg, alcoholic steatohepatitis; drug-induced, viral, or autoimmune hepatitis; primary biliary cirrhosis; primary sclerosing cholangitis; hemochromatosis; alpha 1 antitrypsin deficiency; Wilson's disease) including positive results for hepatitis B surface antigen (HBsAg) or hepatitis C antibody tests (anti-HCV).
3. History of cirrhosis and/or hepatic decompensation, including ascites, hepatic encephalopathy or variceal bleeding.
4. Prior or planned liver transplantation.
5. Alcohol consumption > 21 units of alcohol per week for men and > 14 units per week for women on average over a two-year time frame prior to baseline biopsy.
6. Evidence of alcohol dependence as assessed by the Alcohol Use Disorder Identification Test (AUDIT) questionnaire at screening
7. A history of type 1 diabetes mellitus (T1DM), a history of diabetic ketoacidosis or current use of insulin-based therapies.
8. Clinically significant inflammatory bowel disease or other severe disease or surgery affecting the upper GI tract (including bariatric surgery) which may affect gastric emptying or could affect the interpretation of safety and tolerability data
9. Physician-diagnosed diabetic subjects with clinically significant gastroparesis (as judged by the investigator) or those treated for gastroparesis within 6 months prior to screening
10. History of > 5 kg weight loss in the last 6 months prior to screening or recent (within 3 months of screening) use of drugs approved for weight loss (eg, orlistat, bupropion / naltrexone, phentermine-topiramate, phentermine, lorcaserin), as well as those drugs used off-label.
11. Clinically significant cardiovascular or cerebrovascular disease within the past 3 months, including but not limited to, myocardial infarction, acute coronary syndrome or stroke, or subjects who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening.
12. Severe congestive heart failure (New York Heart Association Class IV).
13. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer.
14. History of substance dependence or a positive screen for drugs of abuse, likely to impact subject safety or compliance with study procedures, at the discretion of the investigator.
15. History of psychosis or bipolar disorder. History of major depressive disorder within the past year with the subject being clinically unstable, or any history of suicide attempt or history of suicidal ideation within the past year.
16. Recent (within 3 months of baseline biopsy) use of therapies associated with development of NAFLD (eg, systemic corticosteroids, methotrexate, tamoxifen, amiodarone, or long-term use of tetracyclines).
17. Recent (within 3 months of baseline biopsy) use of obeticholic acid or other therapy under investigation for NASH.
18. High dose vitamin E (> 400 IU) unless on a stable dose for at least 1 year prior to the baseline biopsy, and not initiated after the biopsy was taken.
19. Recent (within 3 months of baseline biopsy) use of GLP-1 receptor agonist or GLP-1 receptor agonist containing therapies.
20. Any subject who has received another investigational product as part of a clinical study within the last 30 days or 5 half-lives of the therapy (whichever is longer) at the time of screening. Any prior exposure to MEDI0382 is not permitted.
21. Concurrent participation in another interventional study of any kind or repeat randomization in this study.
22. Severe allergy/hypersensitivity to any of the proposed study treatments or excipients.
23. Contra-indication to MRI: such as subjects with pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field; subjects with history of extreme claustrophobia or subject cannot fit inside the MR scanner cavity.
24. History of acute pancreatitis or current chronic pancreatitis. Subjects with serum triglyceride concentrations above 1000 mg/dL (11 mmol/L) at screening, as this can precipitate acute pancreatitis.
25. Abnormal laboratory values including any of the following:

    1. AST or ALT > 5 × ULN.
    2. Impaired renal function defined as estimated glomerular filtration rate (eGFR) ≤ 30 mL/minute/1.73 m2 at screening (estimated according to chronic kidney disease epidemiology collaboration [CKD-EPI]).
    3. Albumin < 35 g/L.
    4. International normalized ratio (INR) > 1.3.
    5. Total Bilirubin (TBL) > 25 µmol/L in the absence of known Gilbert's disease.
    6. Platelets < 140-150,000/mm3
    7. Any other clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the investigator.
26. Severely uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 180 mm Hg and/or diastolic blood pressure (DBP) ≥ 110 mm Hg on the average of 2 seated measurements after being at rest for at least 10 minutes at screening or randomization.
27. Basal calcitonin level > 50 ng/L at screening, or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN 2).
28. Hemoglobinopathy, hemolytic anemia, or chronic anemia (hemoglobin concentration < 11.5 g/dL [115 g/L] for male subjects or < 10.5 g/dL [105 g/L] for female subjects) at screening, or any other condition known to interfere with interpretation of HbA1c measurements
29. Any positive results for human immunodeficiency virus (HIV) infection.
30. Any AstraZeneca, MedImmune, contract research organization (CRO), or study site employee, or close relatives of any of the aforementioned employees.
31. Females who are pregnant or lactating.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (22):
  - Research Site, Tucson, Arizona
  - Research Site, Canoga Park, California
  - Research Site, Chula Vista, California
  - Research Site, Coronado, California
  - Research Site, La Jolla, California
  - Research Site, Lincoln, California
  - Research Site, Los Angeles, California
  - Research Site, Montclair, California
  - Research Site, Torrance, California
  - Research Site, Westminster, California
  - Research Site, Doral, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Marrero, Louisiana
  - Research Site, Las Vegas, Nevada
  - Research Site, Durham, North Carolina
  - Research Site, Blue Ash, Ohio
  - Research Site, Chattanooga, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
- Research Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Shankar SS, Daniels SJ, Robertson D, Sarv J, Sanchez J, Carter D, Jermutus L, Challis B, Sanyal AJ. Safety and Efficacy of Novel Incretin Co-agonist Cotadutide in Biopsy-proven Noncirrhotic MASH With Fibrosis. Clin Gastroenterol Hepatol. 2024 Sep;22(9):1847-1857.e11. doi: 10.1016/j.cgh.2024.04.017. Epub 2024 May 9. PMID 38729399
- See also: d5671c00002-csp-amendment-6 - Redacted - 31Mar2022 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5671C00002&attachmentIdentifier=4696a0aa-270e-46eb-8cd6-cdd51aeab7f9&fileName=d5671c00002-csp-amendment-6_-_Redacted_-_31Mar2022.pdf&versionIdentifier=
- See also: d5671c00002-CSR-synopsis - Redacted - 31Mar2022 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5671C00002&attachmentIdentifier=a7e025dc-807a-4619-91f1-e5cdf18d7fb1&fileName=d5671c00002-CSR-synopsis_-_Redacted_-_31Mar2022.pdf&versionIdentifier=
- See also: d5671c00002-sap-v5 - Redacted - 31Mar2022 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5671C00002&attachmentIdentifier=add9be93-0d96-4b60-8510-b5d6d2ca6d31&fileName=d5671c00002-sap-v5_-_Redacted_-_31Mar2022.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- MEDI0382 300 ug: MEDI0382 300 ug
- MEDI0382 600 ug: MEDI0382 600 ug
- Placebo: Placebo
Period: Overall Study
Arm/Group | MEDI0382 300 ug | MEDI0382 600 ug | Placebo
Started | 25 | 25 | 24
Completed | 21 | 23 | 19
Not Completed | 4 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI0382 300 ug | MEDI0382 600 ug | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 24 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (10.5) | 59.4 (11.9) | 52.2 (13.5) | 55.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 14 | 41
  Male | 13 | 10 | 10 | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 1 | 1
  ASIAN | 0 | 0 | 0 | 0
  BLACK OR AFRICAN AMERICAN | 1 | 1 | 0 | 2
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0 | 0
  WHITE | 24 | 24 | 23 | 71

OUTCOME MEASURES:

1. Primary Outcome: Safety (Including Hepatic Safety) and Tolerability of MEDI0382 Compared With Placebo: Number of Participants With TEAE and SAE
Description: The number and percentage of treatment emergent adverse events (TEAE) and serious adverse events (SAE) through the end of the follow-up period
Time Frame: Day 1 - Day 161
Measure: Count of Participants; unit: Participants
Groups:
- MEDI0382 300ug: MEDI0382 300ug
- MEDI0382 600ug: MEDI0382 600ug
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 26 | 24 | 24
Participants
  Participants with any AE | 20 | 22 | 9
  Participants with any AE with outcome of death | 0 | 0 | 0
  Participants with any SAE (including events with outcome of death) | 1 | 1 | 1
  Participants with any AE leading to discontinuation of investigational product | 2 | 4 | 1
  Participants with any AE leading to withdrawal from study | 0 | 0 | 0

2. Secondary Outcome: Immunogenicity Profile Defined by Presence of Anti-drug Antibodies (ADA): ADA Titer (if Confirmed Positive)
Description: Development of ADA titer (if confirmed positive)
Time Frame: Day 1 - Day 161 (Baseline, Week 6, Week 12, Week 16, Week 19 and Week 23)
Population: Number Analyzed per Row reflects the participants with positive ADA results at each time point. With zero positive ADA results Number Analyzed is zero for Participants.
Measure: Median (Full Range); unit: ADA titer
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 26 | 24 | 24
ADA titer
  Baseline: number analyzed (Participants) | 1 | 0 | 0
  Baseline | 15 [15 to 15] |  |
  Week 6: number analyzed (Participants) | 2 | 1 | 0
  Week 6 | 120 [120 to 120] | 60 [60 to 60] |
  Week 12: number analyzed (Participants) | 8 | 6 | 0
  Week 12 | 30 [15 to 960] | 15 [15 to 30] |
  Week 16: number analyzed (Participants) | 8 | 9 | 0
  Week 16 | 60 [15 to 480] | 60 [15 to 60] |
  Week 19: number analyzed (Participants) | 8 | 9 | 0
  Week 19 | 120 [15 to 480] | 30 [15 to 120] |
  Week 23: number analyzed (Participants) | 7 | 9 | 0
  Week 23 | 120 [15 to 480] | 30 [15 to 240] |

3. Secondary Outcome: Immunogenicity Profile Defined by Presence of Anti-drug Antibodies (ADA): Number of Participants With Development of ADA
Description: Development of ADA during treatment and follow-up
Time Frame: Day 1 - Day 161
Population: As-treated
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 25 | 25 | 24
Participants
  Number of subjects with a positive result at baseline | 1 | 0 | 0
  Number of subjects with a positive result at Week 2: number analyzed (Participants) | 24 | 25 | 21
  Number of subjects with a positive result at Week 2 | 0 | 0 | 0
  Number of subjects with a positive result at Week 6: number analyzed (Participants) | 21 | 23 | 21
  Number of subjects with a positive result at Week 6 | 2 | 1 | 0
  Number of subjects with a positive result at Week 12: number analyzed (Participants) | 20 | 23 | 19
  Number of subjects with a positive result at Week 12 | 8 | 6 | 0
  Number of subjects with a positive result at Week 16: number analyzed (Participants) | 21 | 23 | 18
  Number of subjects with a positive result at Week 16 | 8 | 9 | 0
  Number of subjects with a positive result at Week 19: number analyzed (Participants) | 20 | 21 | 17
  Number of subjects with a positive result at Week 19 | 8 | 9 | 0
  Number of subjects with a positive result at Week 23: number analyzed (Participants) | 19 | 21 | 17
  Number of subjects with a positive result at Week 23 | 7 | 9 | 0

4. Secondary Outcome: Change From Baseline to Week 19 in Hepatic Fat Fraction (HFF)
Description: Change from baseline is defined as the week 19 post-baseline value minus the baseline value. The Analysis of Covariance (ANCOVA) model was used to fit change at week 19. The group of treatment was considered as a fixed effect of the model while the baseline value as covariate. Last observation carried forward (LOCF) method was applied to handle missing data.
Time Frame: Baseline to week 19
Population: The intent-to-treat (ITT) population includes all enrolled participants who are randomized. ITT population was analyzed according to the randomized treatment group. The analyses include those participants who discontinue from study treatments but are still followed up for their scheduled visits.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 21 | 23 | 22
Percent | -1.25 (1.294) | -4.85 (1.236) | 0.16 (1.262)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.439, ANCOVA; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-5.02 to 2.20]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Final Values) = -5.01, 95% CI 2-sided [-8.54 to -1.48]

5. Secondary Outcome: Percent Change From Baseline to Week 19 in Liver Volume
Description: Percent change from baseline is calculated as the week 19 post-baseline value minus the baseline value divided by the baseline value *100. The Analysis of Covariance (ANCOVA) model was used to fit percent change at week 19. The group of treatment was considered as a fixed effect of the model while the baseline value as covariate. Last observation carried forward (LOCF) method was applied to handle missing data.
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 21 | 23 | 22
Percent change | -0.886 (2.7979) | -8.669 (2.6504) | 0.622 (2.6182)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.695, ANCOVA; Mean Difference (Final Values) = -1.508, 95% CI 2-sided [-9.191 to 6.174]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.016, ANCOVA; Mean Difference (Final Values) = -9.291, 95% CI 2-sided [-16.760 to -1.822]

6. Secondary Outcome: Percent Change From Baseline to Week 19 in Liver Fat Volume
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 21 | 23 | 22
Percent change | -2.466 (10.6732) | -29.121 (10.2021) | 8.274 (10.1350)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.468, ANCOVA; Mean Difference (Final Values) = -10.740, 95% CI 2-sided [-40.174 to 18.695]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.012, ANCOVA; Mean Difference (Final Values) = -37.395, 95% CI 2-sided [-66.380 to -8.409]

7. Secondary Outcome: Percent Change From Baseline to Week 19 in Visceral Adipose Tissue
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 18 | 20 | 21
Percent change | 3.359 (3.3107) | -2.152 (2.8958) | -2.901 (2.9198)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.166, ANCOVA; Mean Difference (Final Values) = 6.260, 95% CI 2-sided [-2.698 to 15.218]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.856, ANCOVA; Mean Difference (Final Values) = 0.749, 95% CI 2-sided [-7.537 to 9.035]

8. Secondary Outcome: Percent Change From Baseline to Week 19 in Subcutaneous Adipose Tissue
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 13 | 17 | 15
Percent change | -2.240 (2.4326) | -1.778 (1.8751) | 1.042 (1.9478)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.302, ANCOVA; Mean Difference (Final Values) = -3.283, 95% CI 2-sided [-9.641 to 3.076]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.304, ANCOVA; Mean Difference (Final Values) = -2.821, 95% CI 2-sided [-8.316 to 2.675]

9. Secondary Outcome: Percent Change From Baseline to Week 19 in Liver Diffusion
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 19 | 22 | 20
Percent change | 2.864 (2.9769) | 2.932 (2.7798) | 1.826 (2.9634)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.808, ANCOVA; Mean Difference (Final Values) = 1.038, 95% CI 2-sided [-7.493 to 9.569]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.786, ANCOVA; Mean Difference (Final Values) = 1.106, 95% CI 2-sided [-7.043 to 9.255]

10. Secondary Outcome: Percent Change From Baseline to Week 19 in Abdominal Sagittal Diameter
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 15 | 18 | 17
Percent change | 2.791 (1.4722) | -1.044 (1.2793) | -0.657 (1.2881)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.087, ANCOVA; Mean Difference (Final Values) = 3.448, 95% CI 2-sided [-0.524 to 7.421]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.834, ANCOVA; Mean Difference (Final Values) = -0.387, 95% CI 2-sided [-4.085 to 3.312]

11. Secondary Outcome: Percent Change From Baseline to Week 19 in Abdominal Transversal Diameter
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 15 | 18 | 17
Percent change | 0.605 (0.8585) | -0.100 (0.7458) | 0.991 (0.7443)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.735, ANCOVA; Mean Difference (Final Values) = -0.386, 95% CI 2-sided [-2.681 to 1.908]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.308, ANCOVA; Mean Difference (Final Values) = -1.091, 95% CI 2-sided [-3.226 to 1.044]

12. Secondary Outcome: Percent Change From Baseline to Week 19 in Alanine Aminotransferase (ALT)
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 24 | 24 | 22
Percent change | -10.414 (10.1837) | -15.465 (10.1654) | 8.863 (10.6258)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.195, ANCOVA; Mean Difference (Final Values) = -19.277, 95% CI 2-sided [-48.704 to 10.150]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.103, ANCOVA; Mean Difference (Final Values) = -24.328, 95% CI 2-sided [-53.674 to 5.019]

13. Secondary Outcome: Percent Change From Baseline to Week 19 in Gamma Glutamyl Transferase (GGT)
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 24 | 24 | 22
Percent change | -5.876 (13.6449) | 11.600 (13.6079) | 4.514 (14.2134)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.600, ANCOVA; Mean Difference (Final Values) = -10.390, 95% CI 2-sided [-49.802 to 29.022]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.720, ANCOVA; Mean Difference (Final Values) = 7.086, 95% CI 2-sided [-32.163 to 46.336]

14. Secondary Outcome: Percent Change From Baseline to Week 19 in Aspartate Aminotransferase (AST)
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 24 | 24 | 22
Percent change | -3.447 (9.0121) | -13.951 (8.9326) | 5.693 (9.2942)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.485, ANCOVA; Mean Difference (Final Values) = -9.140, 95% CI 2-sided [-35.134 to 16.854]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.131, ANCOVA; Mean Difference (Final Values) = -19.645, 95% CI 2-sided [-45.288 to 5.999]

15. Secondary Outcome: Percent Change From Baseline to Week 19 in Body Weight
Description: as for outcome 5
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 25 | 25 | 23
Percent change | -1.286 (0.8589) | -2.933 (0.8624) | -0.568 (0.8959)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.564, ANCOVA; Mean Difference (Final Values) = -0.719, 95% CI 2-sided [-3.191 to 1.754]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.062, ANCOVA; Mean Difference (Final Values) = -2.366, 95% CI 2-sided [-4.854 to 0.122]

16. Secondary Outcome: Change From Baseline to Week 19 in Body Mass Index (BMI)
Description: as for outcome 4
Time Frame: Baseline to week 19
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: kg/m2
Arm/Group | MEDI0382 300ug | MEDI0382 600ug | Placebo
Number analyzed (Participants) | 25 | 25 | 23
kg/m2 | -0.349 (0.3200) | -1.042 (0.3202) | -0.265 (0.3338)
Statistical Analysis 1: Comparison: MEDI0382 300ug vs Placebo; Test type: Superiority; p = 0.856, ANCOVA; Mean Difference (Final Values) = -0.084, 95% CI 2-sided [-1.007 to 0.838]
Statistical Analysis 2: Comparison: MEDI0382 600ug vs Placebo; Test type: Superiority; p = 0.098, ANCOVA; Mean Difference (Final Values) = -0.777, 95% CI 2-sided [-1.700 to 0.147]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events and Serious Adverse Events are summarized from the first dose of IP throughout the treatment period of 19 weeks and including the follow-up period of 4 weeks - a total of 23 weeks.
Description: One participant randomized to 600ug received 300ug.
Arm/Group | MEDI0382 300 ug | MEDI0382 600 ug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/24 | 0/24
Other Adverse Events (participants affected / at risk) | 20/26 | 22/24 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI0382 300 ug (N=26) | MEDI0382 600 ug (N=24) | Placebo (N=24)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI0382 300 ug (N=26) | MEDI0382 600 ug (N=24) | Placebo (N=24)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (28) | 20 (42) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 10 (17) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 3 (3) | 1 (1) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Blood calcitonin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 5 (5) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04019561/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04019561/SAP_003.pdf